CLINICAL TRIAL: NCT02683980
Title: Ablation Efficacy of Contact Side Firing Fiber in Predefined Settings for Treating BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-SBU-VP-15-02
Record Dates: First submitted 2016-01-31; First posted 2016-02-17 (Estimated); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Treatment of Benign Prostatic Hyperplasia

ARMS (1):
- Ablation of the prostate (Experimental): ablation of the prostate will be performed using the study device: Lumenis Pulse P120H Holmium Laser
  Interventions: Device: Lumenis Pulse P120H and Xpeeda side firing fiber

INTERVENTIONS:
Device: Lumenis Pulse P120H and Xpeeda side firing fiber

SUMMARY:
Twenty (20) subjects presenting with a hyperplasia enlarged prostate and candidates for surgery will undergo a single treatment for ablation of the prostate using the study device. Follow up visits are scheduled for the day of release from the hospital and at 1 and 3 months post procedure.

The primary objective of this study is to explore Vaporization efficacy and safety when treating BPH (Benign prostatic hyperplasia) with the contact side firing fiber with recommended settings.

ELIGIBILITY:
Inclusion Criteria:

* Subject will be older than 18 years of age
* Subject was diagnosed with enlarged prostate of ≥ 30 gr volume
* Subject is a candidate for surgery treatment
* Subject is willing and has signed the Informed Consent Form
* AUA score ≥ 12
* Qmax <15 mL/s

Exclusion Criteria:

* Need to perform concomitant procedure, other than prostate vaporization
* PVR > 300 mL
* Current Urine retention and Pdet <40 cm H20
* Documented or suspected prostate cancer and / or bladder cancer
* Neurogenic bladder disorder / neurogenic voiding dysfunction
* Urethral strictures
* Previous prostatic, bladder neck, or urethral surgery
* Known history of spinal cord injury
* Urogenital trauma
* Bladder neck stricture
* Evidence of urinary tract infection
* History of chronic prostatitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York Methodist Hospital, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ablation of the Prostate: ablation of the prostate will be performed using the study device: Lumenis Pulse P120H Holmium Laser
  Lumenis Pulse P120H and Xpeeda side firing fiber
Period: Overall Study
Arm/Group | Ablation of the Prostate
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Ablation Time
Description: Calculate the lasing time (in minutes) to ablate the prostate as an indication for treatment efficiency.
Time Frame: Intraprocedural (procedure time is typically 1 to 3 hours)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
Minutes | 36.0 (19.3)

2. Primary Outcome: Ablation Rate
Description: Ablation rate is the change in prostate volume measured by trans-rectal ultrasound divided by the procedure time.
  Ablation rate= (baseline prostate volume - 3-Month prostate volume in mL) / Procedure time in minutes
Time Frame: Baseline and 3-month follow-up visit
Measure: Mean (Standard Deviation); unit: mL/minutes
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
mL/minutes | 0.4 (0.2)

3. Primary Outcome: Efficiency of the Laser to Ablate the Prostate
Description: Ablation efficiency is the change in prostate volume, as measured by trans-urethral ultrasound, between baseline and the 3-month follow-up visit divided by energy.
  Efficiency = (Baseline prostate volume in mL - prostate volume at the 3-month follow-up visit) / energy in J
Time Frame: Baseline and 3-month follow-up visit
Measure: Mean (Standard Deviation); unit: mL/Joules
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
mL/Joules | 9.4 (6.9)

4. Primary Outcome: Safety: Intraoperative Complications
Description: Number and type of intraoperative complications
Time Frame: Intraoperative (procedure time is typically 1 to 3 hours)
Measure: Number; unit: number of events
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
number of events
  Conversion to Transurethral resection procedure (TURP) to complete procedure | 1
  Conversion to TURP to maintain hemostasis | 0
  Capsule perforation | 0
  Bleeding - occurred several times but could be controlled | 3
  Blood transfusion | 0

5. Primary Outcome: Safety: Perioperative Complications
Description: Number of Re-Catheterizations and number of Readmissions were evaluated within this Outcome Measure. Erectile Dysfunction is reported separately. Other complications with reporting of Level of Severity (mild, moderate, or severe) are listed as part of this Outcome Measure. These other complications were Bleeding, Dysuria, Hematuria, Urgency, Urinary Incontinence, Urinary Retention, Frequency, and Nocturia
Time Frame: Post-procedure through 3 months
Population: All patients were assessed post-procedurally through the 3-month follow-up visit for number of Re-Catheterizations, Readmissions and other complications including Bleeding, Dysuria, Hematuria, Urgency, Urinary Incontinence, Urinary Retention, Frequency, and Nocturia.
Measure: Number; unit: Events
Units Other Than Participants: Specific intraoperative complications
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
Number analyzed (Specific intraoperative complications) | 28
Events
  Recatheterization | 2
  Readmission | 0
  Peri-procedure Urinary Retention (mild) | 1
  Urinary retention (mild) at 1 month post procedure | 1
  Urinary retention (moderate) at 1 month post procedure | 1
  Peri-procedure Urgency (mild) | 1
  Urgency (mild) at 1 month | 5
  Urgency (mild) at 3 months | 1
  Urinary Incontinence (mild) at 1 month | 1
  Dysuria (mild) at 1 month | 2
  Dysuria (mild) at 3 months | 1
  Peri-procedure Hematuria (mild) | 2
  Hematuria (mild) at 3 months post procedure | 1
  Bleeding (mild) at hospital discharge | 1
  Bleeding (mild) at 1 month post procedure | 1
  Frequency (mild) 1 month post procedure | 3
  Frequency (mild) 3 months post procedure | 2
  Nocturia (mild) 1 month post procedure | 1
  Nocturia (mild) 3 months post procedure | 1

6. Secondary Outcome: Erectile Dysfunction
Description: Sum score of International Index of Erectile Function (IIEF-5) questionnaire which measures erectile function, orgasmic function, sexual desire, and satisfaction. Each question is ranked 1-5 with a total sum score of 5 (severe erectile dysfunction) to 25 (normal function).
Time Frame: Baseline and 3-month follow-up visit
Population: 19 participants had evaluable data at baseline, and 16 participants had evaluable data from the 3-month follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 19
score on a scale
  Baseline | 6.1 (4.9)
  3-Month Follow-up: number analyzed (Participants) | 16
  3-Month Follow-up | 8.9 (8.5)

7. Secondary Outcome: Visibility During Procedure
Description: Rating on a scale of 1 (Poor) to 5 (Excellent) of the visibility during the procedure
Time Frame: Intraprocedural (procedure time is typically 1 to 3 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
Participants
  Poor | 0
  Fair | 0
  Good | 4
  Very Good | 7
  Excellent | 9

8. Secondary Outcome: Number of Fibers Used During Procedure
Description: Number of fibers used during the BPH procedure
Time Frame: Intraprocedural (procedure time is typically 1 to 3 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
Participants
  1 fiber used | 17
  2 fibers used | 3
  3 fibers used | 0

9. Secondary Outcome: Catheterization Time
Description: Number of days catheter was in place post-ablation of the prostate
Time Frame: Postoperatively through study completion up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
Participants
  4 to 7 days | 3
  8 to 15 days | 16
  Not provided | 1

10. Secondary Outcome: Hospital Stay Duration
Description: Number of days in hospital
Time Frame: Procedure through discharge from hospital (typically 1 day, but measured through end of study up to 3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
Participants
  1 day | 20
  >1 day | 0

11. Secondary Outcome: International Prostate Symptom Score Quality of Life
Description: The International Prostate Symptom Score (IPSS) is an eight-question written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the lower urinary tract symptoms of benign prostatic hyperplasia (BPH). The Quality of Life question has a scale of 0-6, with 0=delighted and 6=terrible.
Time Frame: Baseline, 1-month and 3-month follow-up visits
Population: 20 participants, 17 participants, and 18 participants had evaluable data at baseline, 1-month, and 3-month follow-up visits, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
score on a scale
  Baseline | 3.4 (1.2)
  1-Month Follow-up: number analyzed (Participants) | 17
  1-Month Follow-up | 2.6 (2.2)
  3-Month Follow-up: number analyzed (Participants) | 18
  3-Month Follow-up | 1.9 (2.0)

12. Secondary Outcome: Qmax Uroflow
Description: The maximum urine flow rate (Qmax) is a measure of the quantity of urine excreted in a specified period of time, expressed in cubic centimeters/second (cc/sec).
Time Frame: Baseline, 1-month and 3-month follow-up visits
Population: 20 participants had evaluable data at baseline. 17 participants and 19 participants had evaluable data from the 1-month and 3-month follow-up visits, respectively.
Measure: Mean (Standard Deviation); unit: cc/sec
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
cc/sec
  Baseline | 7.3 (3.9)
  1-month follow-up visit: number analyzed (Participants) | 17
  1-month follow-up visit | 12.8 (6.6)
  3-month follow-up visit: number analyzed (Participants) | 19
  3-month follow-up visit | 9.4 (5.0)

13. Secondary Outcome: PVR (Post-void Residual)
Description: Volume of urine remaining in the bladder after voiding, measured via ultrasound
Time Frame: Baseline, 1-month and 3-month follow-up visits
Population: 20 participants had evaluable data at baseline and the 1-month follow-up visit. 19 participants had evaluable data at the 3-month follow-up visit.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
mL
  Baseline | 63.0 (60.5)
  1-month follow-up visit | 44.9 (31.8)
  3-month follow-up visit: number analyzed (Participants) | 19
  3-month follow-up visit | 55.9 (40.8)

14. Secondary Outcome: PSA (Prostate-specific Antigen)
Description: Prostate-specific antigen, or PSA, is a protein produced by cells of the prostate gland. Prostate cancer can cause elevated PSA levels.
Time Frame: Baseline and 3-month follow-up visit
Population: 15 participants and 19 participants had evaluable data at the baseline and 3-month interval, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 19
ng/mL
  Baseline: number analyzed (Participants) | 15
  Baseline | 2.1 (1.5)
  3-month follow-up visit | 2.1 (1.4)

15. Secondary Outcome: Americal Urological Association (AUA) Symptom Index
Description: The American Urological Association (AUA) Symptom Index assesses the severity of lower urinary tract symptoms in men, particularly related to benign prostatic hyperplasia. The AUA Symptom Score ranges from 0 to 35, with higher scores indicating more severe urinary symptoms related to benign prostatic hyperplasia (BPH).
Time Frame: Baseline, 1-month and 3-month follow-up visits
Population: 20, 17, and 20 participants had evaluable data at baseline, 1-month and 3-month follow-up visits, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ablation of the Prostate
Number analyzed (Participants) | 20
score on a scale
  Baseline | 18.4 (4.3)
  1-month follow-up visit: number analyzed (Participants) | 17
  1-month follow-up visit | 13.8 (9.5)
  3-month follow-up visit | 10.5 (7.4)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Ablation of the Prostate
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 12/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation of the Prostate (N=20)
Urgency (Renal and urinary disorders) | 6 (7)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 3 (3)
Bleeding (Renal and urinary disorders) | 1 (1)
Other (Renal and urinary disorders) | 1 (1) — Frequency, mild
Other (Renal and urinary disorders) | 1 (1) — Mild nocturia
Other (Renal and urinary disorders) | 1 (1) — "Failed TOV POD #1, foley placed easily for outpatient D/C."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT02683980/Prot_SAP_000.pdf